CLINICAL TRIAL: NCT06658327
Title: Comparative Effects Of Dynamic And Static Stretching On Pain, Lower Extremity Function And Knee Range Of Motion In Postmenopausal Females With Knee Osteoarthritis
Brief Title: Comparative Effects Of Dynamic And Static Stretching In Postmenopausal Females With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tanzeela Majeed
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Postmenopausal; Knee Osteoarthritis
Keywords: Pain; Postmenopausal; knee Osteoarthritis; Dynamic Stretching; Static Stretching
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Dynamic stretching
  Interventions: Other: Dynamic stretching
- Group B (Experimental): Static Stretching
  Interventions: Other: Static stretching

INTERVENTIONS:
Other: Dynamic stretching — Group A will receive 2*10 repetitions of dynamic stretching of hamstrings and calf muscles in standing position after application of hot pack (standard size which had been stored in a hydro collator tank of 74.5-80°C for 30 minutes) with 6-8 layers of towel was applied on lower extremity for 10 minutes The subjects will be asked to stand upright with their feet parallel and facing forward with hands holding onto something. Each treatment session will last for 30 minutes. The protocol will be repeated every day for 5 days from the first day of treatment.
  Arms: Group A
Other: Static stretching — Group B will receive 2*10 repetitions of static stretching of hamstrings and quads in standing position after application of hot pack (standard size which had been stored in a hydro collator tank of 74.5-80°C for 30 minutes) with 6-8 layers of towel was applied on lower extremity for 10 minutes. The subjects will be asked to stand upright with their feet parallel and facing forward with hands holding onto something. Each treatment session will last for 30 minutes. The protocol will be repeated every day for 5 days from the first day of treatment.
  Arms: Group B

SUMMARY:
As the aging population continues to grow, there is a pressing need to explore effective interventions to alleviate the symptoms of osteoarthritis, particularly in postmenopausal women who may experience unique challenges. Osteoarthritis (OA) is progressive joint disease characterized by joint inflammation and a reparative bone response and is one of the top five most disabling conditions that affects more than one-third of persons >65 years of age, commonly affecting hands, feet, spine, hips, and knees. Among the various therapeutic modalities, stretching exercises, both dynamic and static, have gained attention for their potential to enhance joint flexibility, reduce pain, and improve functional outcomes.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial and will be conducted in Jinnah Hospital, Mafaza-Tul-Hayat Hospital Lahore and Mayo Hospital Lahore. This study will be completed in time duration of 7 months after the approval of synopsis. Non-probability convenience sampling technique will be used and 58 participants will be recruited in study after randomization. The subjects will be divided into two groups. Group A will receive dynamic stretching of hamstrings and quadriceps with static stretching and Group B will receive dynamic stretching without static stretching after warm up as baseline treatment. The tools that will be used are Osteoarthritis outcome scale Goniometer Lower extremity function scale, Strength, MMT, NPRS, after data collection data will be analyzed by using SPSS version 21

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 65
* Diagnosed patients of OA with grade 3
* Multiparous (5 children)
* Fertile females
* Pain greater than 6 on NPRS

Exclusion Criteria:

* BMI > 30
* Early menarche ≤10 or 11 years.
* Cancer i.e breast cancer ,Ovrian cancer
* Any bone deformity before menopause i.e limb length discrepancy, angulation

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
GONIOMETER | 6 Weeks
  Goniometer is a device used to measure joint ranges. Goniometric measurement of ROM is an important part of clinical examination in osteoarthritis knee and can give information about available knee joint motion, guide about pattern of management, and prognosis.
LOWER EXTREMITY FUNCTION SCALE | 6 Weeks
  The LEFS scores demonstrated excellent test-retest reliability (intraclass correlation coefficients ranging between 0.85 and 0.99) and demonstrated the expected relationships with measures assessing similar constructs.
STRENGTH MMT | 6 Weeks
  MMT is the most commonly used method for documenting impairments in muscle strength. Manual muscle testing is used in rehabilitation and recovery to evaluate contractile units, including muscles and tendons, and their ability to generate forces.
Numerical Pain Rating Scale | 6 Weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tanzeela Majeed, MS, Principal Investigator — Ripah International university, Lahore
Locations (1):
- Mafaza-Tul-Hayat Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Jung JH, Bang CH, Song GG, Kim C, Kim JH, Choi SJ. Knee osteoarthritis and menopausal hormone therapy in postmenopausal women: a nationwide cross-sectional study. Menopause. 2018 Dec 21;26(6):598-602. doi: 10.1097/GME.0000000000001280. PMID 30586007